CLINICAL TRIAL: NCT00398307
Title: A Phase I, Open-Label Study Evaluating the Pharmacokinetics of Components of S-1 in Patients With Varying Degrees of Renal Function
Brief Title: Evaluating Patients With Varying Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1111
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Renal Impairment
Keywords: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — S-1 plus cisplatin

INTERVENTIONS:
Drug: S-1/Cisplatin — S-1 administration will be determined by degree of renal impairment as follows:
  Group A (Control): 30 mg/m2 BID Group B (Mild renal dysfunction): 30 mg/m2 BID Group C (Moderate renal dysfunction): 20 mg/m2 BID Group D (Severe renal dysfunction): 20 mg/m2 QD
  Pharmacokinetic Phase (Part 1):
  On Days -2 and 14 of the Pharmacokinetic Phase, patients will receive a single dose of S-1 administered orally in the morning.
  Treatment will be followed by 1 week of recovery (Days 15 through 21).
  Extension Phase (Part 2):
  S-1 will be administered orally for 2 weeks (Day 1 through Day 14) followed by a 1-week recovery period (Day 15 through Day 21). This cycle will be repeated every 3 weeks.

SUMMARY:
This is a Phase I, open-label study evaluating the PK of S-1 components and their metabolites in patients with advanced solid tumors and varying degrees of renal function. Patients will be stratified by baseline 24-hour creatinine clearance(CrCL) into 4 cohorts using the normal clearance formula:

Group A: Control Group B:Mild renal dysfunction Group C:Moderate renal function and Group D: Severe renal dysfunction. Six patients will be enrolled into each cohort.

ELIGIBILITY:
Inclusion Criteria:

* A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study:

  1. Has histologically or cytologically proven advanced solid tumors for which no standard therapy exists.
  2. Has provided written informed consent.
  3. Is 18 years of age or older.
  4. Is able to take medications orally.
  5. Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to ≤ 2 Appendix A,ECOG Performance Status).
  6. Has adequate organ function as defined by the following criteria:

     1. Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times the upper limit of normal(ULN). If liver function abnormalities are due to underlying malignancy, then AST(SGOT) and ALT (SGPT) may be ≤ 5 times ULN.
     2. Total serum bilirubin ≤ 1.5 times ULN.
     3. Absolute granulocyte count ≥ 1,500/mm3 (ie, ≥ 1.5 x 109/L by International Units [IU]).
     4. Has a platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L).
     5. Has a hemoglobin value of ≥ 9.0 g/dL.
  7. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

3.3.2 Exclusion Criteria

Exclude a patient from this study if he/she does not fulfill the inclusion criteria, or if any of the following conditions are observed:

1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

   1. Any investigational agent received either concurrently or within the last 30 days.
   2. Previous therapy for malignancy within 21 days, including any chemotherapy, immunotherapy, biologic or hormonal therapy (6 weeks for nitrosoureas or mitomycin(C).
   3. Previous radiotherapy within 14 days.
   4. Current enrollment in another clinical trial.
2. Has a serious illness or medical condition(s) including, but not limited to, the following:

   1. Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure (New York Heart Association [NYHA] Class III or IV, Appendix E, NYHA Classification).
   2. Known (at the time of entry) gastrointestinal disorder, including malabsorption, chronic nausea, vomiting, or diarrhea present to the extent that it might interfere with oral intake and absorption of the study medication.
   3. Known brain metastasis.
   4. Known leptomeningeal metastases.
   5. Requires hemodialysis.
   6. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome(AIDS)-related illness.
   7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
3. Is receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

   1. Sorivudine, uracil, dipyridamole, cimetidine and folinic acid (may enhance S-1 activity).
   2. Allopurinol (may diminish S-1 activity).
   3. Phenytoin (S-1 may enhance phenytoin activity).
   4. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 and flucytosine activity).
   5. Pilocarpine (may inhibit CYP2A6 activity).
4. Has known sensitivity to 5-FU.
5. Is a pregnant or lactating female.
6. Is a patient with reproductive potential who refuses to use an adequate means of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To provide specific dosing recommendations for S-1 in patients with renal impairment based on the PK of S-1 and its components after single dose and steady state conditions. | The Pharmacokinetic Phase (Part 1) of the study will last 24 days.

SECONDARY OUTCOMES:
Assess Anti-tumor activity, and safety profile of S-1 in patients with impaired renal function | Each cycle of the Extension Phase (Part 2) will be 21 days (14 days of S-1 treatment, 7 days recovery). The end of study for the Extension Phase will be 30 days after the last dose of S-1.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - LAC/USC Medical Center, Los Angeles, California
  - Premiere Oncology, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Kentucky/Division of Hematology/Oncology and Blood Marrow Transplantation, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cancer Research & Treatment Center/University of New Mexico, Albuquerque, New Mexico
  - The Institute for Drug Development, San Antonio, Texas